CLINICAL TRIAL: NCT06380153
Title: To Evaluate the Pharmacokinetics of Hemay005 Tablets in Subjects With Mild and Moderate Renal Impairment and Normal Renal Function After a Single Oral Administration
Brief Title: To Evaluate the Pharmacokinetics of Hemay005 Tablets in Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM005PS1S07
Record Dates: First submitted 2024-04-09; First posted 2024-04-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Hemay005

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild renal impairment group (Experimental): 15mg/tablet，Four tablets (60mg) each time. Participants will receive a single dose of Hemay005 tablet in Day1
  Interventions: Drug: Hemay005
- Moderate renal impairment group (Experimental): 15mg/tablet，Four tablets (60mg) each time. Participants will receive a single dose of Hemay005 tablet in Day1
  Interventions: Drug: Hemay005
- Healthy subjects (Experimental): 15mg/tablet，Four tablets (60mg) each time. Participants will receive a single dose of Hemay005 tablet in Day1
  Interventions: Drug: Hemay005

INTERVENTIONS:
Drug: Hemay005 — 15mg/tablet，Four tablets (60mg) each time. Participants will receive a single dose of Hemay005 tablet in Day1
  Other Names: Hemay005 tablet

SUMMARY:
The aim of this study was to evaluate the pharmacokinetics of Hemay005 tablets in subjects with mild to moderate renal impairment and normal renal function, and to provide a basis for the formulation of clinical medication regimens for patients with renal impairment.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetics and safety of Hemay 005 tablets in subjects with mild to moderate renal impairment and normal renal function, and to provide a basis for the formulation of clinical medication regimens for patients with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* 1.Fully understand the content, process and possible adverse reactions of the trial before the trial, and be able to complete the study and sign the informed consent according to the requirements of the trial protocol;

  2.adults of both sexes aged 18-70 years old (both ends, whichever is based on written informed consent);

  3. The body weight of male subjects was not less than 50 kg and that of female subjects was not less than 45 kg. Body mass index (BMI) : 19-32 kg/m2 (including cut-off value);

  4.The creatinine clearance rate (CLcr, calculated by Cockcroft-Gault formula) of the subjects met the CKD staging criteria of the corresponding groups, namely mild renal impairment: 60≤CLcr<90 mL/min; Moderate renal impairment: 30≤CLcr<60mL/min. At the same time, according to the investigator's judgment, the creatinine clearance rate of the subjects was not expected to change significantly by the end of the study.

  5. Stable renal function: the interval between two creatinine tests was at least 3 days (30 days before the first test result was acceptable), and the fluctuation value of serum creatinine results between the two tests (calculated by the formula: (the second result-the first result)/the first result) was less than 30%;

  6.no new concomitant medications in the 2 weeks before screening, no adjustment in the treatment regimen (including the type, dose, or frequency of medications) for underlying diseases in the 4 weeks before screening, and no change in the treatment regimen (except for drugs used temporarily on demand) during the study (except as specified in the protocol), or no medication was used;

  7.In addition to renal impairment and complications, the investigators were in good physical condition according to medical history inquiry, vital signs, physical examination, laboratory tests (blood routine, urine routine, stool routine, blood biochemistry, coagulation function, blood pregnancy (only female), 12-lead electrocardiogram, chest X-ray, abdominal color Doppler ultrasound, etc.), and no other clinically significant abnormalities.

Exclusion Criteria:

* 1.(Inquired) The subject has any of the following conditions: acute kidney failure, a history of kidney transplantation, or a need for kidney transplantation or any type of dialysis during the planned trial period; Patients with urinary incontinence or anuria; Patients with obstructive urinary tract diseases (such as urinary tract obstruction caused by urinary calculi, urinary tract obstruction caused by abdominal space occupying lesions, etc.), and the investigator thought that they were not suitable;

  2. (Inquiry) In addition to the disease causing renal impairment, patients with serious acute or chronic diseases of other vital organs within 1 year prior to screening, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, liver, gastrointestinal system, respiratory system, metabolic system, skeletal system and other systems, who were judged by the investigator to be not suitable for the trial;

  3. (Inquiry) Any of the following occurred in the 6 months prior to study entry: Myocardial infarction, Congenital long QT syndrome, Torsades de pointes (including sustained ventricular tachycardia and ventricular fibrillation), right bundle branch block and left anterior hemiblock (bifascicular block), Unstable angina pectoris, coronary artery/peripheral artery bypass grafting, New York Heart Association (NYHA) class III or IV congestive heart failure, cerebrovascular accident, transient ischemic attack, or pulmonary embolism;

  4. (inquiring) patients with a history of depression or suicidal tendencies;

  5. (inquiry) patients who had severe gastrointestinal diseases or had digestive system surgery within 3 months before screening, which affected drug absorption according to the investigator;

  6.(inquiry) blood loss or donation of more than 400mL within one month before screening, or red blood cell transfusion;

  7. Screening laboratory test results met any of the following: (a) alanine aminotransferase (ALT) >2 times the normal value; (b) total bilirubin >1.5 times the normal value; (c) neutrophil count <1.3×109/L; (d) hemoglobin <80g/L; (e) platelet count <80×109/L;

  8.(inquiry) with specific allergic history (asthma, urticaria, eczema, etc.), or allergic condition (such as allergic to two or more drugs, foods or pollens), or known allergic to PDE4 inhibitors (such as apast, roflumilast, etc.);

  9. (queried) drug users in the past 3 years or drug abuse in the past 5 years;

  10. screening positive for drug abuse (excluding those screened positive for drug abuse due to concomitant medications);

  11. with positive breath alcohol test (alcohol concentration >0mg/L);

  12. (inquired) drank more than 14 units of alcohol per week in the 3 months before screening (1 unit = 17.7 mL ethanol, i.e. 1 unit = 354 mL of 5% beer or 44 mL of 40% liquor or 147 mL of 12% wine), or could not abstain from alcohol during the study;

  13.(inquired) smoked more than 5 cigarettes per day in the 3 months before screening, or could not stop using any tobacco products during the study;

  14. (questionnaire) consuming excessive amounts of tea, coffee and/or caffeine-rich beverages (> 8 cups, 1 cup =250 mL) per day in the previous 3 months;

  15. Hepatitis B, hepatitis C, HIV and syphilis tests have one or more clinical significance;

  16. (inquiry) who had participated in and used other drug/device clinical trials within 3 months before screening;

  17. (inquiry) use of any drugs (e.g., inductors-barbiturates, pioglitazone, carbamazepine, phenytoin, glucocorticoids) that induce or inhibit hepatic drug-metabolizing enzymes within 30 days before screening; Inhibitors: SSRI antidepressants, cimetidine, diltiazem macrolides, nitroimidazole, sedative hypnotics, verapamil, fluoroquinolones, antihistamines, isoniazid);

  18. (inquiry) who had used prescription drugs, over-the-counter drugs, health supplements, herbal products or vaccines other than those used to treat renal impairment and other concomitant diseases within 2 weeks before screening;

  19. (inquiry) consumed any caffeine/xanthine/food or drink (such as strong tea, coffee, chocolate, cola, animal organs, grapefruit, dragon fruit, mango, etc.) rich in caffeine/xanthine/which may affect the absorption, distribution, metabolism, and excretion of the drug in the investigator's decision from screening to -1 day of admission, or could not stop consuming the above food or drink during the study;

  20. (inquiry) pregnant or lactating women, or subjects (including male subjects) who have plans to have children or to donate sperm or eggs from two weeks before the study to six months after the last dose of the study, and who are unwilling or unable to use effective contraception;

  21.(inquiry) unable to eat or have swallowing difficulties, have special dietary requirements and/or cannot follow a uniform diet;

  22. (inquiry) with a history of epileptic seizures;

  23. (inquiry) can not tolerate venipuncture and/or have a history of dizziness;

  24.subjects with other factors considered by the investigator to be ineligible for the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Relevant pharmacokinetic parameters，Peak Plasma Concentration（Cmax） | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，Area under the plasma concentration versus time curve（AUC0-t） | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，Area under the curve from time 0 extrapolated to infinite time (AUC0-inf) | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，half-life (T1/2) | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，clearance (CL/F) | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，volume of distribution (Vz/F) | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters ，Renal clearance rate（CLr） | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic

CONTACTS AND LOCATIONS:
Overall Officials: Weiyong Li, Principal Investigator — Study Principal Investigator
Locations (1):
- Union Hospital of Tongji Medical College; Huazhong University of Science and Technology, Wuhan, Hubei, China